CLINICAL TRIAL: NCT00922961
Title: Research for Predictive Biologic Parameters of Cutaneous Hypersensitivity After Brachytherapy in Breast Cancer
Acronym: MAMMOSITE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAMMOSITE2
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: brachytherapy, late cutaneous toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cellular apoptosis (Experimental)
  Interventions: Biological: Blood sample; Procedure: Clinical exam

INTERVENTIONS:
Biological: Blood sample — Blood sample taken for the analysis of the rate of CD8 T-Lymphocyte Apoptosis
Procedure: Clinical exam — Assessment of the esthetic score, and the late cutaneous side effect by 2 physicians

SUMMARY:
25 patients, treated by brachytherapy in a phase II study "Mammosite" (from 2003 to 2005), will be asked to attend a clinical exam in order to evaluate the late cutaneous toxicity due to brachytherapy.

During this consultation, a blood sample will be taken for analysis ( rate of CD8 T-Lymphocyte Apoptosis)

DETAILED DESCRIPTION:
This is an interventional study for the french law

ELIGIBILITY:
Inclusion Criteria:

* All patient treated by exclusive per-operative brachytherapy in the prior study Mammosite for breast cancer
* Patient with social security

Exclusion Criteria:

* Not applicable

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the rate of Radiation-Induced CD8 T-Lymphocyte Apoptosis | Blood sample during a consultation

SECONDARY OUTCOMES:
Assessment of the rate and scores of late fibrosis related to irradiation by mammosite | During a consultation with 2 physicians
Assessment of the rate of telangiectasia | During a consultation with 2 physicians
Assessment of the rate of sequellar pain | During a consultation with 2 physicians
Assessment of the rate of seroma collection | During a consultation with 2 physicians
Assessment of the breast esthetic score | During a consultation with 2 physicians

CONTACTS AND LOCATIONS:
Overall Officials: Yazid BELKACEMI, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France